CLINICAL TRIAL: NCT00479895
Title: Phase II, Open-Label Study in the Catheterization Laboratory Setting to Challenge the Concept That HBOC-201 Administration Might Improve Myocardial 'Oxygenation' and Myocardial Function at the Moment of (Brief) Coronary Occlusion
Brief Title: Hemoglobin Based Oxygen Therapeutics in Elective Percutaneous Coronary Revascularization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biopure Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: COR-0002
Record Dates: First submitted 2007-05-25; First posted 2007-05-28 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Occlusion; Acute Coronary Syndrome
Keywords: Percutaneous Coronary Intervention; Myocardial Ischemia; Balloon Occlusion; Catheter Lab
MeSH Terms: conditions — Coronary Occlusion; Acute Coronary Syndrome; Myocardial Ischemia | interventions — HBOC 201

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Occlusion with pre-oxygenated HBOC-201 followed by dry occlusion
  Interventions: Drug: Hemoglobin Based Oxygen Carrier-201 (HBOC-201, Hemopure)
- 2 (Other): Dry occlusion followed by occlusion with pre-oxygenated HBOC-201
  Interventions: Drug: Hemoglobin Based Oxygen Carrier-201 (HBOC-201, Hemopure)

INTERVENTIONS:
Drug: Hemoglobin Based Oxygen Carrier-201 (HBOC-201, Hemopure) — Pre-oxygenated HBOC-201

SUMMARY:
The test compound and subject of this clinical trial is the haemoglobin-based oxygen carrier, HBOC-201 (Hemopure). HBOC-201, initially developed as an alternative to red blood cells for surgical patients, has the ability to restore tissue oxygenation in persistently ischemic tissue. The development of this new class of compounds, referred to as oxygen therapeutics, provides an opportunity to test the safety and efficacy of a new approach to management of myocardial ischemia.

DETAILED DESCRIPTION:
Because of their ability to perfuse and deliver oxygen, hemoglobin-based oxygen carriers (HBOC) may be considered in the treatment of several ischemic conditions, such as acute coronary syndromes (ACS). Elective percutaneous intervention (PCI) induces transient myocardial ischemia due to reduction of coronary flow during balloon inflation in the coronary artery, thus simulating in a control setting, the occurrence of an ACS.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before initiation of any study-related procedure and agreement to comply with all protocol-specific procedures
* Stable angina pectoris (CCS Class 1, 2, 3, 4) or unstable angina (Braundwald class 1-3, B) or documented silent ischemia
* Baseline ECG with stable sinus rhythm and no signs of ischemia and with no Q waves, bundle branch block or IV conduction disturbances.
* Normal left ventricular wall motion on left ventricular angiogram or on echocardiogram with preserved systolic global LV function
* Non-occlusive stenosis, located in the proximal segments of the left anterior descending artery (LAD) (segments 6 and/or 7) and/or circumflex artery (CFX) (segments 11 and/or 12) or right coronary artery (RCA) (segments 1, 2 and/or 3) for which there is clinical indication to percutaneous treatment with coronary stenting
* Successful PCI with stenting on the target vessel
* Older than 18 years and younger than 80 years of age

Exclusion Criteria:

* Active ischemia at the initiation of the study procedure
* Non-ST segment elevation myocardial infarction
* History or ECG evidence of prior MI in the territory supplied by the vessel undergoing PCI, IV conduction defects/baseline ST-segment abnormalities on the surface ECG
* Moderate to severe aortic or mitral valve disease
* Evidence of LV hypertrophy on the echocardiogram IVS > 13 and/or PW > 13mm
* Angiographically visible collateral vessels to the target vessel
* Hypertension not adequately controlled by anti-hypertensive therapy at the time of study entry (> 140/100mmHg)
* Uncompensated congestive heart failure or signs of pulmonary edema
* Significant hemodynamic compromise and/or cardiogenic shock requiring inotropic or pressor support
* Contraindications to standard drugs for coronary intervention and coronary heart disease: aspirin, heparin, low molecular weight heparin, clopidogrel, contrast dye
* Confirmed pregnancy
* Systemic mastocytosis
* Hypoxemia (need for mechanical ventilation
* Known history of COPD with FEV 1s < 1.0 liter
* Renal impairment: creatinine > 1.6 mg/dl
* Participation in another trial with an investigational drug or device including follow-up period, within the last 30 days before enrollment

Additional exclusion criteria at the end of PCI (before randomization)

* Coronary TIMI flow in the treated artery is less than 3
* Serious arrhythmias during/following the PCI was noted
* Coronary spasm following PCI
* Any deterioration in the subject's "risk" status between informed consent and randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To study the change in left ventricular relaxation indices and pressure-half time and the change in the sum of ST segment deviations compared to baseline. | Duration of the study

SECONDARY OUTCOMES:
LV hemodynamics; change of ST segment; QCA analysis before and after the no-infusion control occlusion and HBOC-201 infusion/occlusion; safety endpoints | Duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: A. Gerson Greenburg, MD, PhD, Study Director — Biopure Corporation
Locations (1):
- Thoraxcentre - Erasmus MC, Rotterdam, Netherlands